CLINICAL TRIAL: NCT00839514
Title: Evaluation of Parkinson Disease Symptoms in Trichloroethylene Exposed Patients in an Industrial Population
Brief Title: Trichloroethylene (TCE) Exposure in an Industrial Population
Acronym: TCE
Status: Completed | Type: Observational
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, John Slevin, Principal investigator, University of Kentucky
Other Study IDs: 08-0301
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Trichloroethylene
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to follow-up with workers from a local company that had exposure to TCE that may have symptoms of Parkinson's disease. We hope to learn more about TCE exposure and Parkinson's disease. Eligible participants will be those who participated in previous research study entitled "Survey of Selected Exposures and Neurologic Symptoms in an Industrial Population"

ELIGIBILITY:
Inclusion Criteria:

* Previous participant in the research study entitled "Survey of Selected Exposures and Neurologic Symptoms in an Industrial Population"

Exclusion Criteria:

* Not a participant in the research study entitled "Survey of Selected Exposures and Neurologic Symptoms in an Industrial Population"

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Follow-up with individuals who previously particpated in the research study entitled "Survey of Selected Exposures and Neurologic Symptoms in an Industrial Population"
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John T Slevin, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Background] Gash DM, Rutland K, Hudson NL, Sullivan PG, Bing G, Cass WA, Pandya JD, Liu M, Choi DY, Hunter RL, Gerhardt GA, Smith CD, Slevin JT, Prince TS. Trichloroethylene: Parkinsonism and complex 1 mitochondrial neurotoxicity. Ann Neurol. 2008 Feb;63(2):184-92. doi: 10.1002/ana.21288. PMID 18157908